CLINICAL TRIAL: NCT03230201
Title: Impact of Lymph Node Dissection in the Management of High-risk Primary Upper Tract Urothelial Carcinoma Patients
Brief Title: Lymph Node Dissection in High-risk UTUC(Upper Tract Urothelial Carcinoma)
Acronym: UTUC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xuesong Li, Professor, Peking University First Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IUPU-16-UTUC-3
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Recurrence; Metastasis; Upper Tract Urothelial Carcinoma; Lymph Node Dissection
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis | interventions — Lymph Node Excision

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blank control (No Intervention): do not receive Lymph node dissection during surgery.
- Lymph node dissection (Experimental): will receive Lymph node dissection during radical nephroureterectomy.
  Interventions: Procedure: Lymph node dissection

INTERVENTIONS:
Procedure: Lymph node dissection — Lymph node dissection during radical nephroureterectomy
  Arms: Lymph node dissection

SUMMARY:
This clinical trial is designed to evaluate the role of lymph node dissection in the prevention of recurrence and metastasis after radical nephroureterectomy for high-risk primary upper tract urothelial carcinoma (UTUC) patients.

DETAILED DESCRIPTION:
INTRODUCTION Upper tract urothelial carcinomas (UTUC) are relatively uncommon compared to bladder cancer and account for only 5-10% of urothelial carcinomas, with an estimated annual incidence in Western countries of

~2 cases per 100,000 inhabitants. The therapeutic role of regional lymph node dissection (LND) for patients with UTUC remains undetermined. Most reports have supported its staging benefit in which patients with no lymph node metastases (pN0) and those with pathological node metastasis (pN+) are stratified from those without LND (pNx). However, the therapeutic benefit of LND remains controversial. This discrepancy might be attributed to two factors. First, there remains a lack of standardization in the extent of LND. Kondo T et al and Matin SF et al previously reported the primary sites of lymphatic metastases from a mapping study, and then determined the anatomical extent of regional lymph nodes. Second, all results reported so far have been, to the best of our knowledge, derived from retrospective studies. Thus, the current guideline recommends LND for invasive UTUC on the basis of insufficient evidence. AIM OF THE WORK This clinical trial is designed to evaluate the role of lymph node dissection in the prevention of recurrence and metastasis after radical nephroureterectomy for high-risk primary upper tract urothelial carcinoma (UTUC) patients. PATIENTS AND METHODS Patients Type of the study: A randomized controlled trial (RCT), phase II. Study locality: Department of Urology, Peking University First Hospital. Institute of Urology, Peking University. National Urological Cancer Center, Beijing, China. Study design: Patients who was ready to receive nephroureterectomy for high-risk primary UTUC will be prospectively randomized into two groups using excel software by random table function. I. Group 1: will receive LND during radical nephroureterectomy. II. Group 2: do not receive LND during surgery.

Inclusion Criteria:

I. Suspected high-risk UTUC patients without metastases in their preoperative radiological imaging (cN0M0).II. Suspected high-risk UTUC patients without history of bladder tumor.

III. Suspected high-risk UTUC patients without synchronous bladder tumor. IV. Suspected high-risk UTUC patients without contralateral UTUCs.

Exclusion criteria:

I. Patients with significant metastases in their preoperative radiological imaging.

II. Patients with history of bladder tumor. III. Patients with synchronous bladder tumor. IV. Patients with contralateral UTUCs. V. Patients with advanced stage (T4). VI. Patients with other malignant tumors. Methods Intervention Patients who sign an informed consent for agreement to participate will be randomly allocated into one of the two groups using excel software by random table function at the day of nephroureterectomy. In group 1, patients will receive LND during radical nephroureterectomy. While for patients in group 2, no LND will be received. All data will be prospectively maintained and include patients' demographics, preoperative laboratory parameters, operative details and postoperative complications Follow up The scheduled follow up will be according to the EAU guidelines (Rouprêt et al., 2015) by scheduling a urine cytology and cystoscopy at 3 months then yearly while CT urography every year for non-invasive tumors and every 6 months over 2 years and then yearly for invasive tumors. All chemotherapy-related complications will be reported. Outcome and end-point The primary outcome of the study is to determine the overall survival (OS). The secondary outcome is to determine the adverse events postoperative morbidity, mortality and other survival (RFS, CSS, EFS) of patients with high-risk UTUC.

ELIGIBILITY:
Inclusion Criteria:

* I. Suspected high-risk UTUC patients without metastases in their preoperative radiological imaging (cN0M0).II. Suspected high-risk UTUC patients without history of bladder tumor.

III. Suspected high-risk UTUC patients without synchronous bladder tumor. IV. Suspected high-risk UTUC patients without contralateral UTUCs

Exclusion Criteria:

* I. Patients with significant metastases in their preoperative radiological imaging.

II. Patients with history of bladder tumor. III. Patients with synchronous bladder tumor. IV. Patients with contralateral UTUCs. V. Patients with advanced stage (T4). VI. Patients with other malignant tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | three years after surgery

SECONDARY OUTCOMES:
postoperative morbidity and mortality | three years after surgery
recurrence-free survival | three years after surgery
cancer specific survival | three years after surgery
event-free survival | three years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Zhou, M.D., Study Chair — Peking University First Hosipital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China